CLINICAL TRIAL: NCT02641548
Title: Silicone Sock as Treatment of Deep Heel Fissures in People With Diabetes -a Randomized Controlled Trial
Brief Title: Silicone Sock as Treatment of Deep Heel Fissures in People With Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to difficulties in recruiting participants
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Gustav Jarl, PhD, Certified Prosthetist and Orthotist, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OLL-524811
Record Dates: First submitted 2015-12-23; First posted 2015-12-29 (Estimated); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Complications
Keywords: Diabetic foot; Diabetic foot disease; Skin fissures; Xerosis
MeSH Terms: conditions — Diabetes Complications; Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silicone sock+heel cream (Experimental): Every evening a cream (Footmender, Auxilum Cura Innovatio, Dublin, Ireland, European Patent 2522342) is applied to the feet and a sock of silicone is used every night.
  Interventions: Device: Sock of silicone; Other: Heel cream
- Heel cream (Active Comparator): Every evening a cream (Footmender, Auxilum Cura Innovatio, Dublin, Ireland, European Patent 2522342) is applied to the feet
  Interventions: Other: Heel cream

INTERVENTIONS:
Device: Sock of silicone
  Arms: Silicone sock+heel cream
Other: Heel cream
  Other Names: Footmender

SUMMARY:
This study evaluates the addition of using a sock of silicone to using a heel cream, in the treatment of heel fissures in people with diabetes, aiming at healing the fissures and preventing them from developing into ulcers. Half of the participants will use the silicone sock and a heel cream, the other half will use the cream only.

DETAILED DESCRIPTION:
Dry skin and heel fissures are common complications of diabetes and can develop into hard-to-heal ulcers that eventually can make amputation of the foot necessary.

Patients are advised to use heel creams to heal fissures and prevent them from developing into ulcers. Clinical observations have suggested that wearing a silicone sock nighttime can heal fissures, but the additional advantage of using a silicone sock compared to use a heel cream only has not been investigated.

Participants will be randomized to an intervention group (silicone sock and heel cream) or a control group (heel cream only) and the healing of fissures and development of new ulcers will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes diagnosis, and
2. Deep heel fissures

Exclusion Criteria:

Factors associated with increased risk of complications:

1. known allergy or hypersensitivity to silicone or ingredients in cream
2. other skin conditions that make use of sock or cream inappropriate
3. strongly fluctuating foot edema
4. ulcer in part of the foot that the sock is in contact with
5. inability of participant or assisting person to handle the silicone sock correctly including daily cleaning.

Factors associated with increased risk that complications are not discovered or reported, such as, dementia, language or other communication impairments, intellectual disability or known substance abuse, AND there is no other person who can provide adequate support to the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Proportion of healing of deep heel fissures | Once every 4 weeks for approx. 6 months
  Heel fissures are defined as fissures involving the dermis. Participants visit a podiatrist who take a photograph later judged by a blinded assessor: presence or absence of deep fissures.
Time to healing of deep heel fissures | Once every 4 weeks for approx. 6 months
  A survival analysis is conducted on the same variable as above.

SECONDARY OUTCOMES:
Severity of skin dryness | Once every 4 weeks for approx. 6 months
  The photographs taken by the podiatrist will be judged by a blinded assessor according to the cracks/fissure item from the Specified symptom sum score (SRRC) instrument.
Number of participants for whom the fissures develop into ulcers | Once every 4 weeks for approx. 6 months
  The presence of ulcers is judged by the podiatrist at the visits.
Number of participants with complications | Once every 4 weeks for approx. 6 months
  The podiatrist fills in a protocol at each visit, documenting observed complications from the heel cream or silicone sock, such as skin redness, and asks the participants for experienced complications, such as, stings when applying the cream.

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Jarl, PhD, Principal Investigator — Region Örebro County, Örebro, Sweden
Locations (1):
- Örebro University Hospital, Örebro, Örebro County, Sweden

IPD SHARING:
Plan to Share IPD: No
Only group level data will be published

REFERENCES:
- [Background] Pham HT, Exelbert L, Segal-Owens AC, Veves A. A prospective, randomized, controlled double-blind study of a moisturizer for xerosis of the feet in patients with diabetes. Ostomy Wound Manage. 2002 May;48(5):30-6. PMID 12046488
- [Background] Bakker K, Apelqvist J, Schaper NC; International Working Group on Diabetic Foot Editorial Board. Practical guidelines on the management and prevention of the diabetic foot 2011. Diabetes Metab Res Rev. 2012 Feb;28 Suppl 1:225-31. doi: 10.1002/dmrr.2253. No abstract available. PMID 22271742
- [Background] Kang BC, Kim YE, Kim YJ, Chang MJ, Choi HD, Li K, Shin WG. Optimizing EEMCO guidance for the assessment of dry skin (xerosis) for pharmacies. Skin Res Technol. 2014 Feb;20(1):87-91. doi: 10.1111/srt.12089. Epub 2013 Jul 2. PMID 23815476
- [Background] Oe M, Sanada H, Nagase T, Minematsu T, Ohashi Y, Kadono T, Ueki K, Kadowaki T. Factors associated with deep foot fissures in diabetic patients: a cross-sectional observational study. Int J Nurs Stud. 2012 Jun;49(6):739-46. doi: 10.1016/j.ijnurstu.2012.01.007. Epub 2012 Feb 14. PMID 22341798